CLINICAL TRIAL: NCT05358379
Title: A Phase 1/2, Open-label, Multicenter Study to Investigate the Safety, Pharmacokinetics, and Efficacy of CYC140, an Oral PLK1 Inhibitor, in Subjects With Advanced Solid Tumors and Lymphoma
Brief Title: A Study to Investigate CYC140, in Subjects With Advanced Solid Tumors and Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cyclacel Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CYC140-101
Record Dates: First submitted 2022-04-19; First posted 2022-05-03 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor, Adult Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: Dose escalation in Phase 1 part
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): Phase 1 = CYC140 administered orally in escalating doses starting at 5mg QD M-F week 1 to 3 for 3 weeks of a 4 week cycle. Subsequent cohorts will escalate in dose and schedule until optimized phase 2 dose and schedule is achieved.
  Interventions: Drug: CYC140
- Phase 2 (Experimental): Phase 2 = Recommended CYC140 phase 2 dose and schedule administered orally in 28-day cycles.
  Interventions: Drug: CYC140

INTERVENTIONS:
Drug: CYC140 — CYC140 is a highly selective, orally- and intravenously- available, ATP-competitive inhibitor of PLK1.

SUMMARY:
This is a 2-part, phase 1/2, open-label, multicenter study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, pharmacogenomics, and efficacy of CYC140 administered orally daily. This study consists of Phase 1 and Phase 2 components in subjects with advanced solid tumors and lymphoma who have progressed despite having standard therapy or for which no standard therapy exists.

DETAILED DESCRIPTION:
Phase 1 part of the study will consist of a dose-escalation and a dose-finding component.

Phase 2 will enroll subjects with locally advanced, recurrent, or metastatic, histologically confirmed advanced solid tumors or lymphoma, who have failed all standard therapies or for whom standard therapy does not exist, into 8 groups:

Group 1: Bladder cancer

Group 2: Breast cancer: Triple-negative breast cancer (TNBC)

Group 3: Lung cancer (non-small cell lung cancer [NSCLC] and small cell lung cancer [SCLC])

Group 4: Hepatocellular carcinoma (HCC) and biliary tract cancer (BTC)

Group 5: Metastatic colorectal cancer (mCRC) including KRAS-mutated mCRC

Group 6: B-cell lymphoma including diffuse large B-cell lymphoma (DLBCL)

Group 7: T-cell lymphoma (cutaneous T-cell lymphoma [CTCL] and peripheral T-cell lymphoma [PTCL])

Group 8: Basket cohort: tumor types that are suspected to have a related mechanism of action but are not included in previous groups including, esophageal, prostate, ovarian and pancreatic cancers

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged ≥ 18 years.
2. Subjects with histological- or cytological-confirmed, advanced cancer who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists

   1. For Phase 1, all tumor types may be enrolled
   2. For Phase 2, subjects will be enrolled as per the study design section above
3. ECOG performance status of 0-2.
4. Subjects who relapsed post-autologous or post-allogeneic transplant are eligible. Post-transplant subjects must be without active fungal disease or significant acute graft-versus-host disease
5. Women of childbearing potential (WOCBP) must have a negative pregnancy test (urine or serum) within 7 days prior to starting the study drug. Both males and females must agree to use effective birth control during the study (prior to the first dose and for 6 months after the last dose) if conception is possible during this interval.
6. Subjects must be able to swallow and retain orally administered medication and not have any clinically significant GI abnormalities that may alter the absorption, such as malabsorption syndrome or major resection of the stomach or bowels.
7. Able to agree to and sign the informed consent and to comply with the protocol.

Exclusion Criteria:

1. Subjects with a history of brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases. Subjects with treated brain metastases that are asymptomatic and have been clinically stable for at least 4 weeks will be eligible.
2. Subjects who have not received vaccines for severe acute respiratory syndrome-corona virus-2 (SARS-COV-2) and have suspected signs and symptoms of the novel coronavirus infection (COVID-19) or have confirmed COVID-19.
3. Subjects with a history of another primary malignancy, other than:

   1. In situ carcinomas, e.g., breast, cervix, and prostate
   2. Locally excised nonmelanoma skin cancer
   3. No evidence of disease from another primary cancer for 2 or more years and has not taken any anti-cancer treatment in 2 years.
4. Any other clinically significant acute or chronic medical or psychiatric condition or any laboratory abnormality that may increase the risk associated with study drug administration or may interfere with the interpretation of study results.
5. Diseases that significantly affect GI absorption of CYC140.
6. Subjects who have impaired cardiac function or clinically significant cardiac disease.
7. Presence of active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment
8. Presence of an active infection requiring intravenous antibiotics
9. Presence of known history of human immunodeficiency virus-1/2 with uncontrolled viral load and on medications that may interfere with metabolism
10. Presence of active hepatitis B virus (HBV) or hepatitis C virus (HCV).
11. Chemotherapy, biologic therapy, targeted therapy, immunotherapy, extended-field radiotherapy, or investigational agents within 5 half-lives or 3 weeks (whichever is shorter) prior to administration of first dose of study drug on Day 1 or have not recovered from the side effects of such therapy.
12. Major surgery/surgical therapy for any cause within 4 weeks of the first dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | 6 months
  The incidence rate of dose-limiting toxicities (first cycle only) at each dose level
Overall Response Rate (ORR) | 18 months
  Assessment of response criteria according to RESIST, Lugano or mSWAT.

SECONDARY OUTCOMES:
Adverse events | 24 months
  Type, frequency, and severity of adverse drug reactions
AUC | 6 months
  CYC140 plasma concentrations
Cmax | 6 months
  CYC140 plasma concentrations
Tmax | 6 months
  CYC140 plasma concentrations
T1/2 | 6 months
  CYC140 plasma concentrations
Disease Control Rate | 24 months
  To evaluate the disease control rate (DCR) in subjects receiving CYC140.
Duration of Response | 24 months
  To evaluate the duration of response (DOR) in subjects receiving CYC140.
Progression-free Survival | 24 months
  To evaluate progression-free survival (PFS) in subjects receiving CYC140.
Overall Survival | 24 months
  To evaluate overall survival (OS) in subjects receiving CYC140.

OTHER OUTCOMES:
Pharmacodynamics | 6 months
  Pharmacodynamic response to CYC140 will be assessed by mRNA sequencing of blood samples to determine differential expression of PLK1 target genes (including MYC, PLK1, CDKN1A) relative to baseline.
Pharmacogenomics | 24 months
  Genomic alterations will be assessed by next generation sequencing (NGS) at baseline and various time points during treatment with CYC140 in order to investigate the relationship between genetic alterations in CYC140 related pathways and response to CYC140.
  Parameters of genetic variations (DNA mutations) and copy number variations using plasma cell-free DNA derived from peripheral blood will be assessed.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (3):
  - City of Hope, Duarte, California
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Seoul National University Hospital, Seoul, South Korea
- Hospital Universitario Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No